CLINICAL TRIAL: NCT04738279
Title: A Study to Determine the Efficacy of Continuous Ambulatory Wearable Technology and a Cascading Alert System in Reducing 30d Readmission in High Risk Heart Failure Patients
Brief Title: The CASCADE HF Soft Launch and Calibration Phase I and II
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Endeavor Health (Other)
Collaborators: physIQ, Inc. (Industry); Carnegie Mellon University (Other); Northwestern University (Other)
Responsible Party: Principal Investigator, Nirav Shah, Medical Director of Quality Innovation and Clinical Practice Analytics, Program Director of Outcomes Research for Quality and Transformation, Endeavor Health
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: EH20-288 Cascade Soft Launch
Record Dates: First submitted 2021-01-27; First posted 2021-02-04 (Actual); Results first posted 2023-02-16 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Phase I: Soft Launch (120 days) (Experimental): The study will conduct a soft launch on the first five HF patients enrolled to finetune process and protocol.
  Interventions: Device: Non-Invasive Continuous Remote Patient Monitoring; Other: Affective Analysis of Participant Response to Continuous Remote Patient Monitoring
- Phase II: Calibration (210 days) (Experimental): After learning from the soft launch and updating the protocol, the study will continue to enroll 15 HF patients for calibration purposes
  Interventions: Device: Non-Invasive Continuous Remote Patient Monitoring; Other: Affective Analysis of Participant Response to Continuous Remote Patient Monitoring

INTERVENTIONS:
Device: Non-Invasive Continuous Remote Patient Monitoring — Continuous remote patient monitoring will consist of continuous collection of physiological data and patient status through a non-invasive wearable solution, connected to a structured cascading escalation management pathway
Other: Affective Analysis of Participant Response to Continuous Remote Patient Monitoring — Survey and qualitative interviewing of participants

SUMMARY:
Invasive telemonitoring has shown promising results in reducing readmissions and health service utilization, and improving patient outcomes; however, such evidence is lacking for non-invasive telemonitoring. Our proposal is to deploy a wearable solution that predicts physiological perturbation comparable to invasive devices and to perform continuous remote patient monitoring; this will be connected to a structured, cascading, escalation pathway involving home health nurses, advanced practitioner providers, specialists, and surgeons, and has the potential to transform care management in the post-discharge period, where patients are the most vulnerable for readmission.

ELIGIBILITY:
Inclusion Criteria:

* Patient is an inpatient at NorthShore University HealthSystem
* Patient is on the heart failure consult list
* Patient has a history of heart failure
* Patient received at least one dose of IV diuretics at index hospitalization
* Patient is discharging with NorthShore Home Health services
* Symptoms corresponding to New York Heart Association function class II-IV
* Patient has heart failure with reduced left ventricular ejection fraction (LVEF)<40%, or HF with mid-ranged ejection fraction (LVEF 40-50%), or HF with preserved ejection fraction (LVEF≥50%)
* Patient is in the top 50% risk of readmission across NorthShore University HealthSystem's CAPE 30-day readmission model
* Patient is at least 18 years of age
* Patient is fluent in English
* Patient agrees to protocol-required procedures

Exclusion Criteria:

* Patient has cognitive or physical limitations that, in the opinion of the investigator, limit the patient's ability to maintain patch, phone
* Patient has allergy to hydrocolloid adhesives
* Patient has present skin damage preventing them from wearing a study device
* Patient has renal dysfunction requiring dialysis
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nirav S Shah, MD, MPH, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University HealthSystem Evanston Hospital, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted at Evanston Hospital during December 2020 to October 2021
Period: Overall Study
Arm/Group | Phase I: Soft Launch (120 Days) | Phase II: Calibration (210 Days)
Started | 5 | 15
Completed | 4 | 13
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I: Soft Launch (120 Days) | Phase II: Calibration (210 Days) | Total
Number analyzed (Participants) | 5 | 15 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 5 | 7
  >=65 years | 3 | 10 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 1 | 11 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 5 | 14 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 12 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Attrition Rate
Description: Drop out from study
Time Frame: 30 days from patient discharge date
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Soft Launch (120 Days) | Phase II: Calibration (210 Days)
Number analyzed (Participants) | 5 | 15
Participants | 1 | 2

2. Primary Outcome: Enrollment Rate
Description: Enrollment rate for entire patient cohort
Time Frame: Through study completion, an average of 30 days for each patient
Population: Overall number of participants analyzed reflects the number of participants who were screened for phase I and phase II, respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Soft Launch (120 Days) | Phase II: Calibration (210 Days)
Number analyzed (Participants) | 43 | 431
Participants | 5 | 15

3. Secondary Outcome: Number of Participants With Diuretic Escalation
Description: Frequency of augmenting diuretic dosage as prescribed by the cardiologist to the patient.
Time Frame: 30 days from patient discharge date
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Soft Launch (120 Days) | Phase II: Calibration (210 Days)
Number analyzed (Participants) | 5 | 15
Participants | 2 | 9

4. Secondary Outcome: 30-day Readmission
Description: 30-day readmission to hospital
Time Frame: 30 days from patient discharge date
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Soft Launch (120 Days) | Phase II: Calibration (210 Days)
Number analyzed (Participants) | 5 | 15
Participants | 2 | 2

ADVERSE EVENTS:
Time Frame: We collected adverse event data over the 30-day participation period for each participant
Arm/Group | Phase I: Soft Launch (120 Days) | Phase II: Calibration (210 Days)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/15
Other Adverse Events (participants affected / at risk) | 0/5 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2022-07-12): https://cdn.clinicaltrials.gov/large-docs/79/NCT04738279/Prot_000.pdf